CLINICAL TRIAL: NCT03147794
Title: Functional Electrical Stimulation Therapy for Children With Upper Limb Weakness Post Stroke: Evaluation of the Mynd Move Technology
Brief Title: Functional Electrical Stimulation for Children With Upper Limb Weakness Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: MyndTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FES Study
Record Dates: First submitted 2017-04-12; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Hemiparesis; Stroke
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES using MyndMove Technology (Experimental): This is the only arm of the study. Participants will be provided with the FES intervention as part of the protocol.
  Interventions: Device: MyndMove

INTERVENTIONS:
Device: MyndMove — A new technology system called MyndMove has been developed by MyndTec Inc. (Missisauga Canada) to administer FES. The purpose of this technology is to improve voluntary upper limb (hand and arm) function (i.e. reaching and grasping) for patients with hemiparesis as a results of stroke or spinal cord injury (7). It is a non-invasive application that delivers electrical stimulation to the affected limb transcutaneously. MyndMove has been licensed by Health Canada and is indicated as a functional electrical stimulator for improvement of arm and hand function and active range of motion in patients with hemiplegia due to stroke or upper limb paralysis due to C3-C7 spinal cord injury.

SUMMARY:
A new technology system called MyndMove has been developed by MyndTec Inc. (Missisauga Canada) to administer FES. The purpose of this technology is to improve voluntary upper limb (hand and arm) function (i.e. reaching and grasping) for patients with hemiparesis as a results of stroke or spinal cord injury (7). It is a non-invasive application that delivers electrical stimulation to the affected limb transcutaneously. MyndMove has been licensed by Health Canada and is indicated as a functional electrical stimulator for improvement of arm and hand function and active range of motion in patients with hemiplegia due to stroke or upper limb paralysis due to C3-C7 spinal cord injury. In a randomized controlled trial looking at adults with acute stroke and limited or complete immobility of the arm, FES and intensive therapy was shown to have significant improvement of hand function compared to the control group that was exposed to intensive therapy only (8). Limited research using MyndMove to administer FES has been conducted for pediatric populations, however there is significant potential for FES and intensive therapy to improve hand function for children with upper extremity hemiparesis using MyndMove technology. Before the efficacy of MyndMove therapy can be evaluated in children age 3 to 6, the tolerability of the system must first be evaluated and proven for this age group.

DETAILED DESCRIPTION:
Research Questions and Objectives:

The overall goal of this study is to determine if therapy administered using MyndMove can be tolerated by children age 3 to 6 with upper extremity hemiparesis and produce effective response without injury or pain.

The objectives of this study are:

1. To evaluate the tolerability of MyndMove technology to safely provide Functional Electrical Stimulation (FES) transdermally as therapy in young children

   From these findings the researchers aim to:
2. To establish clinical recommendations for the next step of this study, which will evaluate the efficacy of MyndMove therapy with this population using a pre-post case series model .

Specifically, this study will answer the following research questions:

1) Can MyndMove FES stimulation be tolerated by young children ages 3 to 6 with upper extremity hemiparesis without pain or discomfort? he following of directions and understanding of the nature of the therapy.

Intervention All participants in this study will receive transcutaneous functional electrical stimulation via MyndMove administered by trained occupational therapists (OTs) from the Acquired Brain Injury department at Holland Bloorview Kids Rehabilitation Hospital. The MyndMove system is a neuromodulation device that delivers short electrical pulses to stimulate muscle contractions and enhance motor recovery following stroke or spinal cord injury. MyndMove delivers therapeutic stimulation sequences called protocols, which are coded therapeutic algorithms which assist muscle contractions for arm and hand movement allowing the brain and central nervous system to be retrained, restoring voluntary reaching and grasping functions lost following neurological injury. The MyndMove system comprises the hardware device, stimulation electrodes and cables, hand and foot switches, and integrated software. OTs will be trained at a 2-day course that trains users on the MyndMove system. The purpose of the workshop is to train users how to safely and effectively use the system, screen for contraindications, and identify eligible clients for MyndMove. OTs will receive instructions on available training protocol and the application of the protocol. The course also includes a practical component, focusing on establishing user's comfort with the MyndMove system (see Appendix 9 for the MyndMove Course Training Outline).

FES will be delivered while participants engage in task-oriented activities that require reaching and grasping. Neuromuscular recover in stroke patients typically starts with recovery of proximal parts and then recovery of distal parts. Therefore, the research team will test tolerability proximally to distally in the protocol. The participant will be asked to perform three to five of the following movements: 1) touch nose, 2) touch opposite shoulder, 3) touch forehead, 4) move arm forward, 5) lift affected arm up and extend elbow, 6) hand opening, 7) palmar grasp, 8) pinch grasp, 9) lateral pinch grasp, and 10) lumbrical grasp. In long-term therapeutic FES interventions, once participants are able to voluntarily control these shoulder and elbow movements, the OT would proceed to focus on the distal parts of the arm. However, because this is a tolerability study and FES will only be administered in one session, the OTs will test the distal parts of the arm even if the participant has not achieved voluntary control of their shoulder and elbow movements. The participants will be asked to perform each specific task for an interval of 10 to 20 seconds. Participants will repeat each task 10 or more times, or as long as the one hour session allows. This session will involve the parent and a child life specialist to increase the child's acceptance during the therapy and to assist in the process of detecting and mitigating discomfort during sessions. Observations will be recorded by the OT as in Part 1. During and after the session, the OT will look for signs and symptoms of discomfort.

ELIGIBILITY:
Inclusion Criteria:

i) Ischaemic or Haemorrhagic stroke with hemiparesis of the upper extremity; ii) Willing to attend therapy; and iii) Communicate effectively in English.

Exclusion Criteria:

i) Global aphasia; ii) Upper extremity condition that limits the function of the hand and arm before the stroke; iii) Active seizure disorder within 5 years; iv) Implanted pacemaker, vagal nerve stimulator, AICD, baclofen pump, or similar implanted metallic or electronic device; v) Unhealed fracture or wound in the affected arm; vi) BOTOX injection into the affected arm or hand within 6 months; vii) Currently enrolled in another study of upper limb therapy or new investigational drugs/biologics within 6 months; viii) Swollen, infected or inflamed areas or skin eruptions on the affected arm including evidence of phlebitis or venous incompetence in the arm; ix) Known cardiac dysrhythmia; x) cancerous or suspected cancerous lesions present on the affected arm and xi) Cognitive impairment sufficient enough to impede in the following of directions and understanding of the nature of the therapy, xii) Unwilling/unable to assent to study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Scale | Administered at Appointment 2 (Day 7 of study)
  This is a pain scale.The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst".

SECONDARY OUTCOMES:
Quality of Upper Extremity Skills Test (QUEST) | Administered at appointment 1 (Day 0 of study)
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rumney, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No
The researchers will not make individual patient data available to other researchers.